CLINICAL TRIAL: NCT00717717
Title: Physical Activity After Cancer Treatment (PACT)- A Clinical Controlled Trial on the Effect of a One-year Physical Activity Program for Cancer Patients Following Cytostatic Treatment
Brief Title: A Clinical Controlled Trial on the Effect of Physical Activity After Cancer Treatment (PACT)
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Velux Fonden (Other); Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Julie Midtgaard, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PACT
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Cancer
Keywords: Cancer Survivor; Physical Activity; Health Behavior; Psychosocial Well-being; Coaching; Long Term; Consequences; Chemotherapy; Motivation
MeSH Terms: conditions — Neoplasms; Motor Activity; Health Behavior | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): No intervention except repeated measurements of physical capacity
- Intervention (Experimental): Intervention: One-year rehabilitation program including weekly supervised and group-based physical exercise, home-based physical activity, individual and group-based coaching (narrative therapy), and expert educational talks/lectures
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — One-year rehabilitation program including weekly supervised and group-based physical exercise, home-based physical activity, individual and group-based coaching (narrative therapy), and expert educational talks/lectures
  Arms: Intervention

SUMMARY:
The PACT Study (Physical Activity after Cancer Treatment) is a unique study within the field of cancer rehabilitation in Denmark. It differs from other studies mainly due to the intervention itself. A combination of physiological, health educational and therapeutic elements will be tested. These components are incorporated into a one-year training program for mixed groups (i.e. men + women, with varying cancer diagnoses) to encourage them to enhance their well.-being and quality of life. The overall aim of this approach is to place increased focus on the treated cancer patient's introduction to and exploitation of both physiological and psychosocial yields through physical exercise. Whether or not the study results bear a positive effect, they are expected to support new knowledge in rehabilitation for cancer survivors.

DETAILED DESCRIPTION:
The PACT ('Physical Activity after Cancer Treatment') Study is a multidisciplinary collaborative study carried out by the University Hospitals Centre for Nursing and Care Research (UCSF) and the Finsen Center (Oncology and Hematology Clinics) of the Copenhagen University Hospital (Rigshospitalet), Copenhagen, Denmark. The project draws in cancer patients who have undergone chemotherapy and who are now disease-free or at a stable phase in their illness and have good prognoses.

The aim of the study is to investigate the effect of a 12-month rehabilitation program comprising supervised and structured physical exercise training (body conditioning; strength-building; relaxation; massage), patient education and coaching combined with a home-based physical exercise group component and will include a control group. Groups of 12-15 patients will be formed (mixed genders; different oncological and hematological diagnoses) who will train together once weekly during the intervention period. Participation in a training program with peers is seen as a positive motivational factor that stimulates and challenges the patient through physical activity, to use his/her own resources to establish sustainable coping strategies.

ELIGIBILITY:
Inclusion Criteria:

* Cancer diagnosis
* Completed cytostatic treatment <6 months
* Affiliated with either the Oncology or Hematology Clinic at the Copenhagen University Hospital, Copenhagen
* Between the ages of 15-70 years
* No evidence of disease or life expectancy >2 years.

Exclusion Criteria:

* Contraindications for physical activity
* Bone and brain metastases
* Multiple myeloma (in the case of hematological patients)
* Symptomatic cardiac illness, including clinical congestive heart disease, treatment caused arrhythmia or myocardial infarction experienced within the previous three months
* Dementia and/or psychosis
* Patients who cannot read or write Danish.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2006-11; Primary Completion 2010-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Physical fitness (VO2Max) | Baseline and follow-up (6, 12, 18, 24, and 36 months)

SECONDARY OUTCOMES:
Muscle strength (1RM) Cholesterol Quality of Life (cancer specific and health related) Anxiety & Depression Fatigue Coping Physical Activity behavior Health Behavior | Baseline and follow-up (6,12,18,24, and 36 months)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Midtgaard, PhD, Principal Investigator — The University Hospitals Centre for Nursing and Care Research (UCSF) / Copenhagen University Hospital (Rigshospitalet); Mikael Rørth, PhD, Study Director — Department of Oncology, Copenhagen University Hospital; Lis Adamsen, Professor, Study Director — The University Hospitals Centre for Nursing and Care Research (UCSF) / Copenhagen University Hospital

REFERENCES:
- See also: Official institutional website — http://www.ucsf.dk